CLINICAL TRIAL: NCT01676415
Title: Role of Short Term Systemic Corticosteroid Therapy in the Management of Chronic Rhinosinusitis Without Nasal Polyps
Brief Title: Corticosteroid Therapy for Chronic Rhinosinusitis Without Nasal Polyps (CRSsNP)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: participants are no longer receiving intervention due to clinical logistics
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Bruce Tan, MD, Assistant Professor, Dept of Otolaryngology, Northwestern University Feinberg School of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18369
Record Dates: First submitted 2012-08-24; First posted 2012-08-30 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Chronic Rhinosinusitis Without Nasal Polyps
Keywords: Sinus disease; Sinonasal complaints; Chronic sinusitis; Nasal polyps; Chronic rhinosinusitis without nasal polyps; Glucocorticoids; Prednisone; Topical mometasone; Anti-inflammatory agents
MeSH Terms: conditions — Paranasal Sinus Diseases; Nasal Polyps | interventions — Prednisone; Glucocorticoids; Mometasone Furoate

ARMS (2):
- Prednisone (Active Comparator): Oral steroid medication
  Interventions: Drug: Prednisone
- Topical Mometasone (Active Comparator): Topical steroid medication
  Interventions: Drug: Topical mometasone

INTERVENTIONS:
Drug: Prednisone — Three-week course of a broad-spectrum antibiotic Amoxicillin/Clavulanate at a daily dosage of 875mg twice daily
  If the subject is allergic to Penicillin and its derivatives or has had an adverse reaction to Amoxicillin/Clavulanate, a three-week course of clarithromycin instead
  Antihistamines if an appropriate history of atopy is obtained
  Systemic prednisone: Starting dose of 40mg for five days followed by a taper decreasing by 10mg every 5 days
  Following completion of the oral corticosteroid: Course of topical mometasone until the end of the study
  Other Names: Glucocorticoid; Deltasone; Liquid Pred; Meticorten; Orasone; Prednicen-M; Prednicot; Sterapred; Sterapred DS
  Arms: Prednisone
Drug: Topical mometasone — Three-week course of a broad-spectrum antibiotic Amoxicillin/Clavulanate at a daily dosage of 875mg twice daily
  If the subject is allergic to Penicillin and its derivatives or has had an adverse reaction to Amoxicillin/Clavulanate, a three-week course of clarithromycin instead
  Antihistamines if an appropriate history of atopy is obtained
  Standing course of topical mometasone at the standard dose of 2 sprays to each nostril once daily and will remain on the topical mometasone until the end of the study.
  Arms: Topical Mometasone

SUMMARY:
The purpose of this study is to determine the most effective route to administer steroids to patients with chronic sinusitis, specifically a type of chronic sinusitis not associated with nasal polyps (CRSsNP). The investigators would like to better understand whether orally administered steroids results in superior results when compared with nasally sprayed steroids. The investigators propose to test the hypothesis that for patients with radiographically proven CRSsNP, routine medical therapy consisting of a short course of systemic corticosteroids is superior to topical corticosteroids for relieving inflammation and the symptoms of CRS.

DETAILED DESCRIPTION:
Chronic sinus infections (chronic sinusitis or CRS) are common conditions that affect millions of Americans. While this is a common disorder, medical treatments for this condition vary a lot and little is known how and why different treatments work in some individuals and not in others. Some physicians commonly utilize a course of oral steroid therapy similar to treatment of inflammatory conditions including asthma and arthritis. Other physicians feel that oral steroids are not more effective than nasal steroid sprays in reducing inflammation and prefer prescribing nasal steroids. There is no conclusive data as to whether oral or sprayed nasal steroids are more effective in providing long-term benefit to patients. Nasal steroids are FDA approved to treat some types of chronic sinusitis but oral steroids are FDA approved medications that are used to treat inflammatory conditions but is not specifically indicated for chronic sinusitis and thus should be regarded as investigational drug. The purpose of this research study is to better understand whether orally administered steroids results in superior results when compared with nasally sprayed steroids. The investigators will compare patients with chronic sinusitis who are first treated with antibiotics and oral steroids, and compare them to chronic sinusitis patients who receive antibiotics and nasally sprayed steroid therapy.

ELIGIBILITY:
Inclusion Criteria:

1. They have three-months of persistent symptoms meeting criteria for chronic rhinosinusitis as defined by the Taskforce on Rhinosinusitis.
2. They have a CT-scan in our clinic or have a viewable recent (< 3weeks prior to clinic visit) CT-scan with a Lund Mckay score of 6 or greater. A Lund Mckay score of 6 or greater is felt to be indicative of at least moderate CRS.
3. They do not have nasal polyps on initial clinic nasal endoscopy
4. They are willing to participate in a clinical study
5. They are between the ages of 18 to 80.

Exclusion Criteria:

1. They have a condition in which the use of systemic corticosteroids is contraindicated such as diabetes will be excluded.
2. They are unable to or unwilling to take the prescribed antibiotics or steroids will excluded.
3. They have been treated with a > 3 week course of antibiotics and/or systemic steroids will also be excluded.
4. They have variants of chronic sinusitis known to be refractory to medical therapy such as Wegener's granulomatosis, primary ciliary dyskinesia or sarcoidosis.
5. They have sinusitis secondary to prior surgery, a dental procedure or anatomical variants.
6. They have nasal polyps on physical exam.
7. They are pregnant. Subjects who are possibly pregnant will be excluded based on history. Pregnancy testing is not standard of care for diagnostic imaging.
8. They have a Lund-Mckay score on CT scan of < 6
9. They are < 18 or > 80 years old

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-08; Primary Completion 2016-01 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Tan, MD, Principal Investigator — Northwestern University
Locations (1):
- : Northwestern Medical Faculty Foundation (NMFF) Sinus and Allergy Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Hissaria P, Smith W, Wormald PJ, Taylor J, Vadas M, Gillis D, Kette F. Short course of systemic corticosteroids in sinonasal polyposis: a double-blind, randomized, placebo-controlled trial with evaluation of outcome measures. J Allergy Clin Immunol. 2006 Jul;118(1):128-33. doi: 10.1016/j.jaci.2006.03.012. Epub 2006 May 19. PMID 16815148
- [Background] Hopkins C, Browne JP, Slack R, Lund V, Brown P. The Lund-Mackay staging system for chronic rhinosinusitis: how is it used and what does it predict? Otolaryngol Head Neck Surg. 2007 Oct;137(4):555-61. doi: 10.1016/j.otohns.2007.02.004. PMID 17903570
- [Background] Hopkins C, Gillett S, Slack R, Lund VJ, Browne JP. Psychometric validity of the 22-item Sinonasal Outcome Test. Clin Otolaryngol. 2009 Oct;34(5):447-54. doi: 10.1111/j.1749-4486.2009.01995.x. PMID 19793277
- [Background] Parikh A, Scadding GK, Darby Y, Baker RC. Topical corticosteroids in chronic rhinosinusitis: a randomized, double-blind, placebo-controlled trial using fluticasone propionate aqueous nasal spray. Rhinology. 2001 Jun;39(2):75-9. PMID 11486442
- [Background] Stankiewicz JA, Chow JM. Cost analysis in the diagnosis of chronic rhinosinusitis. Am J Rhinol. 2003 May-Jun;17(3):139-42. PMID 12862401
- [Background] Wallwork B, Coman W, Mackay-Sim A, Greiff L, Cervin A. A double-blind, randomized, placebo-controlled trial of macrolide in the treatment of chronic rhinosinusitis. Laryngoscope. 2006 Feb;116(2):189-93. doi: 10.1097/01.mlg.0000191560.53555.08. PMID 16467702
- See also: Related Info — http://www.northwestern-sinus.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study had difficult accruing sufficient numbers of patients. Additional Institutional Review Board mandated testing for potential participants made study flow challenging. Study was closed for failure to accrue sufficient patients.
Groups:
- Prednisone: Oral steroid medication
  Prednisone: Three-week course of a broad-spectrum antibiotic Amoxicillin/Clavulanate at a daily dosage of 875mg twice daily
  If the subject is allergic to Penicillin and its derivatives or has had an adverse reaction to Amoxicillin/Clavulanate, a three-week course of clarithromycin instead
  Antihistamines if an appropriate history of atopy is obtained
  Systemic prednisone: Starting dose of 40mg for five days followed by a taper decreasing by 10mg every 5 days
  Following completion of the oral corticosteroid: Course of topical mometasone until the end of the study
- Topical Mometasone: Topical steroid medication
  Topical mometasone: Three-week course of a broad-spectrum antibiotic Amoxicillin/Clavulanate at a daily dosage of 875mg twice daily
  If the subject is allergic to Penicillin and its derivatives or has had an adverse reaction to Amoxicillin/Clavulanate, a three-week course of clarithromycin instead
  Antihistamines if an appropriate history of atopy is obtained
  Standing course of topical mometasone at the standard dose of 2 sprays to each nostril once daily and will remain on the topical mometasone until the end of the study.
Period: Overall Study
Arm/Group | Prednisone | Topical Mometasone
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prednisone | Topical Mometasone | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (16.5) | 45.9 (11.5) | 46.3 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: SNOT-22 Questionnaire
Description: The Sino-nasal Outcome Test-22 is a validated questionnaire that measures 22 nasal and quality of life symptoms ("nasal obstruction" and "loss of smell and taste") ranked from 0 (not a problem) to 5 (problem as bad as it can be).
  Min score= 0, Max score= 110 ("worst possible problem" on all symptoms)
  Change from baseline of the SNOT-22 score. The SNOT-22 questionnaire is a 22-item disease-specific health related quality of life instrument validated for use in chronic rhinosinusitis.
Time Frame: 4-6 weeks and 3 months after initiation of treatment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Prednisone | Topical Mometasone
Number analyzed (Participants) | 4 | 5
units on a scale
  4-6 WEEKS | 45.75 (6.7) | 34.4 (6.0)
  3 MONTHS | 49 (9.3) | 34.4 (8.36)

2. Secondary Outcome: Lund-McKay Score From CT Scan
Description: Change from baseline in Lund-McKay scores from sinus CT-scans at 4-6 weeks and 3 months after initiation of treatment will be used to calculate the overall level of inflammation within the paranasal sinuses.
Time Frame: 4-6 weeks and 3 months after initiation of treatment
Population: Only a few of the patients were able to return for the follow up CT scan, therefore this measure was not analyzed.
Arm/Group | Prednisone | Topical Mometasone
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Taskforce Symptom Inventory
Description: Change from baseline in individual symptom severity. The taskforce symptom inventory is a visual analog scale of the severity of the 4 major symptoms making up the clinical diagnostic criteria of CRS.
Time Frame: 4-6 weeks and 3 months after initiation of treatment
Population: Study had difficult accruing sufficient numbers of patients. Additional Institutional Review Board mandated testing for potential participants made study flow challenging. Study was closed for failure to accrue sufficient patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisone | Topical Mometasone
Number analyzed (Participants) | 4 | 5
Participants | 0 | 0

4. Secondary Outcome: Medication Side-effect and Compliance Inventory
Description: The medication side-effect and compliance inventory is a questionnaire to evaluate the frequency and severity of common side effects associated with the medications used in this study.
Time Frame: 4-6 weeks and 3 months after initiation of treatment
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisone | Topical Mometasone
Number analyzed (Participants) | 4 | 5
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 3 months that patients were enrolled in the study.
Description: The definition of adverse events/serious adverse events do not differ from the Clinical Trials definition. None of the patients in this study had an adverse event or serious adverse event.
Arm/Group | Prednisone | Topical Mometasone
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

LIMITATIONS AND CAVEATS:
Study had difficult accruing sufficient numbers of patients. Additional Institutional Review Board mandated testing for potential participants made study flow challenging. Study was closed for failure to accrue sufficient patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No